CLINICAL TRIAL: NCT04576858
Title: Clinical Utility of Circulating Tumor DNA in Gastro-Esophageal Cancer
Acronym: CURE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Morten Mau-Sørensen, Chief Physician, MD, PhD, Rigshospitalet, Denmark
Other Study IDs: CURE
Record Dates: First submitted 2020-01-23; First posted 2020-10-06 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-09

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: Circulating Tumor DNA
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Cohort 1: Surgical resection + perioperative chemotherapy
  Interventions: Diagnostic Test: Circulating tumor DNA
- Cohort 2: Neoadjuvant chemoradiotherapy followed by surgery
  Interventions: Diagnostic Test: Circulating tumor DNA
- Cohort 3: Definitive chemoradiotherapy
  Interventions: Diagnostic Test: Circulating tumor DNA
- Cohort 4: Chemotherapy with the aim to prolong life expectancy
  Interventions: Diagnostic Test: Circulating tumor DNA
- Cohort 5: Non-chemotherapeutic palliation: E.g. Palliative radiotherapy

INTERVENTIONS:
Diagnostic Test: Circulating tumor DNA — Measurement of circulating tumor DNA from plasma over a period of 2 years.
  Groups: Cohort 1: Surgical resection + perioperative chemotherapy; Cohort 2: Neoadjuvant chemoradiotherapy followed by surgery; Cohort 3: Definitive chemoradiotherapy; Cohort 4: Chemotherapy with the aim to prolong life expectancy

SUMMARY:
This is a prospective cohort study designed to evaluate the treatment effect as well as predictive and prognostic factors with special emphasis on the clinical utility of ctDNA in plasma in patients with gastroesophageal cancer. Patients with gastroesophageal cancer are included in 5 separate cohorts scheduled for

* Surgical resection + perioperative chemotherapy (cohort 1)
* Neoadjuvant chemoradiotherapy followed by surgical resection (cohort 2)
* Definitive chemoradiotherapy with curative intent (cohort 3)
* Systemic therapy with the intent to prolong survival (cohort 4)
* Palliative treatment without the use of chemotherapy (cohort 5)

ELIGIBILITY:
Inclusion Criteria:

Gastroesophageal cancer Age 18 years or older Able to understand and sign written informed consent

Exclusion Criteria:

Patients not providing informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population includes patients with gastroesophageal cancer in five prospective cohorts. Neither WGS/WES on primary tumor nor serial blood samples for ctDNA are mandatory for inclusion in the study. However, it is highly encouraged to perform WGS/WES of the primary tumor. A retrospective cohort will be open for inclusion to facilitate initial hypothesis testing to be validated in the prospective cohorts
Sampling Method: Non-Probability Sample
Enrollment: 1950 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Time to recurrence | 1 year

SECONDARY OUTCOMES:
Time to progression | 1 year
Overall survival | 5 year
Response rate RECIST 1.1 | through study completion, an average of 1 year
Response duration RECIST 1.1 | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark